CLINICAL TRIAL: NCT05636527
Title: A Non-Randomized, Prospective or Retrospective, Open-Label, Multi-Center, Observational Clinical Study With Two Arms to Further Evaluate Safety and Performance of the NEXUS® Aortic Arch Stent Graft System and the Custom-Made NEXUS Multibranch™ Aortic Arch Stent Graft System
Brief Title: Further Evaluation of Safety and Performance of the NEXUS Aortic Arch Stent Graft System and the Custom-Made NEXUS Multibranch™ Aortic Arch Stent Graft System
Acronym: ARCUS
Status: Recruiting | Type: Observational
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP010
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: AAT9

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NEXUS Aortic Arch Stent Graft System
- Custom-made NEXUS Multibranch™ Aortic Arch Stent Graft System

SUMMARY:
The goal of this observational study is to collect clinical information on how safe, and how well the NEXUS Aortic Arch Stent Graft System and the Custom-Made NEXUS DUO™ Aortic Arch Stent Graft System work for the treatment of aortic aneurysms, in the standard-of-care setting.

The main question[s] it aims to answer are:

* Early mortality
* Safety outcomes throughout the study
* Device failure throughout the study
* Procedural and hospitalisation information Participants will be treated per institutional standard of care Follow-up information will be collected through to five years.

ELIGIBILITY:
1. Male and female age ≥18 years
2. The subject is indicated for implant of the NEXUS Aortic Arch System in accordance with the current IFU, or
3. The subject is indicated for implant of the custom-made NEXUS DUO Aortic Arch System in accordance with the current IFU, or
4. The subject has been already implanted, after February 2019, with the NEXUS or the NEXUS DUO according to the relevant IFU
5. The subject is able and willing to provide informed consent to participate in the study.
6. Subject is not currently enrolled in another investigational study or registry that would directly interfere with the current study, except if the subject is participating in a mandatory government registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.
7. In the opinion of the Investigator, life expectancy exceeds one year
8. The subject is not pregnant or planning to become pregnant.
9. In the physician's opinion, subject's renal function is stable for the NEXUS procedure.
10. In the opinion of the investigator, subject does not have co-morbidities or planned surgeries that will interfere with the implant of the device, e.g., major cardiac surgery or interventional procedure in the last 90 days, MI or cerebral vascular accident (CVA) in the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a thoracic aortic aneurysm or chronic dissection extending to or involving the aortic arch and who are considered candidates for the endovascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  The primary outcome in this study is early mortality, defined as lesion related death or any death that occurs within 30-days post-procedure or within initial hospitalization following the index procedure (whichever occurs last), unless there is evidence of accidental or self-inflicted death

SECONDARY OUTCOMES:
Mortality | 12 months
  All-cause death events will be counted
Major Adverse Event (MAE) | 30 days and 12 months
  Occurrence of at least one of the following MAEs at 30 days and 1 year post NEXUS implantation
  * Disabling Stroke
  * Permanent Paralysis/Paraplegia
  * Renal failure
  * Aortic rupture
  * Development of new dissections in the thoracic aorta or brachiocephalic artery
Device failure | Procedure, 30 days, 12 months
  Device Failure will be assessed via the following outcomes:
  * Peri-operative device failure
  * Device occlusion
  * Surgical conversion
  * Re-Intervention to treat migration,
  * Re-Intervention to treat stenosis or occlusion,
  * Re-Intervention to treat type Ia, Ib, III, IV endoleaks
  * Re-Intervention for loss of device integrity

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Schelzig, MD, Principal Investigator — University Hospital Duesseldorf, University Clinic for Vascular and Endovascular Surgery; Augusto D'Onofrio, Principal Investigator — Department of Cardiac, Thoracic, Vascular Sciences and Public Health, University of Padua
Locations (18):
- Belgium (2):
  - Cliniques universitaires Saint Luc, Brussels
  - UZ Leuven, Leuven
- Aretaieio Hospital, Nicosia, Cyprus, Cyprus
- France (2):
  - APHP Henri Mondor, Paris
  - Hôpital Européen Georges Pompidou, Paris
- Germany (4):
  - Immanuel Klinikum Brandenburg, Herzzentrum Brandenburg, Bernau bei Berlin, Brandenburg
  - University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - German Heart Center, Berlin
  - University Hospital Bonn, Bonn
- Evaggelismos General Hospital, Athens, Greece
- Italy (2):
  - Azienda Socio Sanitaria Territoriale (A.S.S.T.) degli Spedali Civili di Brescia, Brescia
  - University Hospital Padoua, Padua
- Netherlands (2):
  - Stichting Amsterdam UMC,, Amsterdam
  - University Medical Center Groningen, Groningen
- Medical University of Warsaw, Warsaw, Poland
- Spain (2):
  - Hospital Universitario Puerta del Mar, Cadiz, Andalusia
  - Hospital Alvaro Cunqueiro Vigo, Vigo, Galicia
- Klinikum Hirslanden, Aorten -und Gefäßzentrum, Zuerich, Zurich, Switzerland